CLINICAL TRIAL: NCT05525845
Title: Physiological Regulation of Energy Intake - The FOOD-PRINT Study Identifying the Hormonal and Neural Footprints of the Visceroceptive, Homeostatic, and Hedonic Components of Food Intake Regulation in Humans
Brief Title: Studying the Hedonic and Homeostatic Regulation of Food Intake Using Functional MRI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Andres J. Acosta, M.D., Ph.D., Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 21-010514
Record Dates: First submitted 2022-08-16; First posted 2022-09-02 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Healthy
MeSH Terms: interventions — immunoglobulin B

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Food-Print Main Arm (Other): Functional Magnetic Resonance Imaging (pCASL-MRI) after Caloric and Volumetric stimulus in lean patients will be performed on all patients in the study
  Interventions: Other: Functional Magnetic Resonance Imaging (pCASL-MRI); Other: Intragastric Balloon; Other: Elemental Meal; Other: Hedonic Meal

INTERVENTIONS:
Other: Functional Magnetic Resonance Imaging (pCASL-MRI) — MRI's will be performed at multiple points on each visit day.
Other: Intragastric Balloon — Intragastric Balloon will be placed during Visit 2 study day and inflated to maximum tolerated volume. Patient will then be scanned in the MRI.
  Other Names: IGB
Other: Elemental Meal — Patient will ingest the tasteless elemental meal until their maximum level of fullness. Once full, the patient will be scanned in the MRI.
Other: Hedonic Meal — Patient will ingest meal of their choice from a local food delivery service and eat until they reach their maximum level of fullness. Once full, the patient will be scanned in the MRI

SUMMARY:
The purpose of this study is to investigate how gut hormones and brain areas respond differently to gastric distention, tasteless calories, or palatable food and how this alters appetite.

ELIGIBILITY:
Inclusion Criteria:

* BMI 18-25 kg/m^2.
* Weight stable for 3 months prior to study entry.
* For females: study days will be scheduled during the follicular phase of their menstrual cycle (i.e., the first 13 days (about 2 weeks) of the cycle).
* Able to provide written informed consent prior to any study procedures and be willing and able to follow study procedures..
* Ability to perform light to moderate physical activity.

Exclusion Criteria:

* Any contraindication for MRI scanning.
* Any history of childhood (> 95th percentile) or adult obesity (BMI >30 kg/m^2).
* Claustrophobia.
* High intensity training or physical activity.
* Any contraindication for intragastric balloon insertion.
* Any allergies to the study meals.
* Any history of eating disorder.
* Any substance abuse disorder (including alcohol and tobacco).
* Any history of psychiatric disorders.
* Any cardiovascular, endocrine, pulmonary, neurological, or gastrointestinal comorbidities.
* Pregnancy or nursing.
* Any history of bariatric surgery or endoscopic bariatric procedure.
* Use of any medication or supplement that alters appetite.
* Patient has a known history of any condition or factor judged by the investigator to prevent participation in the study or which might hinder study adherence.

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2022-09-08 (Actual); Primary Completion 2028-08 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Difference in Cerebral Blood Flow related to hypothalamus | 1 month
  The mean difference in cerebral blood flow (CBF) at fullness (satiation) and return to hunger (satiety) to the hypothalamic area.

SECONDARY OUTCOMES:
Cerebral Bloodflow related in multiple brain areas | 1 month
  The mean difference in cerebral blood flow (CBF) at fullness (satiation) and return to hunger (satiety) to the other brain areas related to food intake regulation.
Cerebral Blood Flow between three stimuli | 1 month
  The mean difference in cerebral blood flow (CBF) between the 3 different stimuli.
Hormone level | 1 month
  Differences in hormones levels (ghrelin, GLP-1, CCK, PYY, leptin, insulin, GIP, amylin) at each of the stages (I.e., baseline, fullness, maximal fullness) after the three different stimulations. These hormones will be compared before and after the same stimulation days. The hormone measurements on stimulation days will also be compared to each other.
comparison of calories | 1 month
  Correlation the caloric consumption to fullness, maximal fullness with degree of cerebral blood flow(CBF) change on PASL MRI.
calorie corellation to hormones | 1 month
  Correlation the caloric consumption to fullness, maximal fullness with changes in the hormonal levels (ghrelin, GLP-1, CCK, PYY, leptin, insulin, GIP, amylin).
hormone level comparison | 1 month
  Differences in the hormonal levels (ghrelin, GLP-1, CCK, PYY, leptin, insulin, GIP, amylin) between fullness and hunger after the three different stimulations. These hormones will be compared before and after the same stimulation days. The hormone measurements on stimulation days will also be compared to each other.
Time differences in stimuli | 1 month
  Differences in time to next meal after maximal fullness after the three different stimulations.
Caloric consumption differences in stimuli | 1 month
  Differences in the caloric consumption after maximal fullness after the three different stimulations.
FitBit measured Physical Activity | 1 month
  Measurement of daily physical activity during free-living conditions measured through the use of FitBit tracker over the duration of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Andres Acosta, MD, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials